CLINICAL TRIAL: NCT03581890
Title: Is Socioeconomic Position Associated With Acute Onset of Colon Cancer and 1-year Mortality After Acute Colon Cancer Surgery
Brief Title: Socioeconomic Position in Acute Colorectal Cancer Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-41-3726
Record Dates: First submitted 2018-03-22; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Neoplasms Malignant
Keywords: Colorectal cancer; Socioeconomic position
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Danish Colorectal Cancer Group (DCCG.dk) database: The DCCG.dk database is a national population-based, clinical database with a completeness proportion of 99% of all colorectal cancer patients in Denmark. Patients are included in the database if treated for or diagnosed with colorectal cancer at a public surgical department in Denmark. No patients underwent treatment for colorectal cancer at private hospitals in Denmark. Metachronous cancers, recurrence, and tumors of other histological origin than primary adenocarcinoma, mucinous adenocarcinoma, signet ring cell carcinoma, medullary carcinoma, or undifferentiated carcinoma are not registered in the DCCG.dk database. The surgeon prospectively registers perioperative variables such as surgical priority, stent insertion and type of colectomy, and patient related variables. Information on postoperative mortality is imported to the database from the Danish Central Civil Registration Registry linking all Danish residents with a unique identification number.
  Interventions: Other: Socioeconomic position

INTERVENTIONS:
Other: Socioeconomic position — Socioeconomic position is the exposure in both study 1 and 2. Four different socioeconomic measures will be tested. The primary socioeconomic position measure is highest attained education the year before surgery (short/medium/long). Secondary measures are:
  1. age- and sex-adjusted available income the year before surgery
  2. Cohabitation status at the year of surgery (living alone/living with a partner) at the year of surgery.
  3. Urbanicity (in four officially, predefined categories).

SUMMARY:
Acute colon cancer surgery has a poor 90-day mortality of 21.0% compared with only 3% after elective colorectal cancer surgery in Denmark. The high mortality after acute colon cancer surgery compared with elective surgery emphasizes the importance of identifying factors associated with acute onset and poor short-term survival after acute surgery. Socioeconomic position has previously showed to be a risk factor for acute versus elective onset of colorectal cancer. Furthermore, if patients with low socioeconomic position have higher postoperative mortality this could reflect differences in the treatment of patients according to their socioeconomic position.

The aim of the clinical study is:

1. To examine if patients with short education, low income, living alone, or living in rural areas are more likely to undergo acute colorectal cancer surgery than elective surgery compared with patients with longer educations, higher income, living with a partner, or living in urban areas.
2. To examine if there is an association between education, income, cohabitation, or urbanicity and 1-year mortality after acute colorectal cancer surgery.

DETAILED DESCRIPTION:
Hypothesis

The investigators hypothesize that patients with short education, low income, living alone, or living in rural areas are, themselves or their physician, less likely to react to unspecified symptoms of colon cancer and have a higher risk of acute onset due to more progressed disease compared with patients with a higher socioeconomic position. Furthermore, the hypothesis is that there is an association between socioeconomic position and 90-day mortality after acute colorectal surgery, explained by patient, treatment or organizational related factors.

Methods

The study is a nationwide, historical cohort study with prospective collected data. All patients in Denmark will be followed up one year after surgery. Exposure is socioeconomic position measured by highest attained education, age and sex-adjusted income, cohabitation status, and urbanicity. Primary outcome in the first study is acute surgical procedure for colorectal cancer. Primary outcome in the second study is year mortality after acute colorectal cancer surgery or insertion of self-expanding metallic stent (SEMS).

Analysis

First study:

Differences in socioeconomic position between patients undergoing acute and elective CRC surgery will be explored with a logistic regression model. We will include the following covariates in the analysis:

Confounders: age, sex.

Mediators: comorbidity (Charlson Comorbidity Index), BMI (Body Mass Index), alcohol, UICC-stage (The Union for International Cancer Control), smoking, tumor localization, income, education, cohabitation, urbanicity A sensitivity analysis will be conducted to examine if department volume adds to the effect of urbanicity.

Second study:

Differences in socioeconomic position in postoperative 1-year mortality after acute colorectal cancer surgery will be analysed with a cox regression model. We will include the following covariates in the analysis:

Confounders: age, sex.

Mediators: comorbidity (Charlson Comorbidity Index), BMI (Body Mass Index), alcohol, UICC-stage (The Union for International Cancer Control), smoking, tumor localization, income, education, cohabitation, urbanicity A sensitivity analysis will be conducted to examine if department volume adds to the effect of urbanicity.

Ethical considerations

The project has been approved by the Danish Data Protection Agency with journal no. 2015-41- 3726. Data will be handled according to Danish law and the Helsinki declaration. This study does not require written content from the participants, thus all data is retracted from databases and registries.

In the presentation of final results all patients will remain anonymous and not identifiable according to Danish law. All data will be kept a minimum of 5 years.

ELIGIBILITY:
Inclusion criteria:

First study

* All patients undergoing a surgical procedure for colorectal cancer in Denmark and registered in the Danish Colorectal Cancer Group (DCCG.dk) database from 1st of January 2007 to 31st of December 2016. If a patient dies during surgery, they will also be included.

Second study

* All patients operated for acute colorectal cancer in Denmark from 1st of January 2007 to 31st of December 2016 and registered in the DCCG.dk database. Acute surgery can either be colectomy, placement of self-expanding metallic stent, diverting stoma, or damage control surgery. If a patient dies during surgery, they will also be included.

Exclusion criteria:

Both studies:

* Not registered In the DCCG.dk database with a colorectal cancer diagnose.
* Missing on income, urbanicity, cohabitation, or UICC-stage.

Second study:

* Registered in the DCCG.dk database with an elective surgical procedure without a registration of SEMS or diverting stoma 72 hours before an emergency admission in NPR.
* lost to follow-up one year postoperative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is retracted from the Danish Colorectal Cancer Group (DCCG.dk) database. See description of the database in cohort description.
  Information regarding highest attained education, age- and sex-adjusted income, cohabitation, and urbanicity will be collected from the registry of education and knowledge, registry of labor, income and wealth, and registry of living conditions via Statistics Denmark, which are nation-wide register with information on health, income, education, family status and other social data from all Danish citizens.
  From the National Patient Registry we collect data regarding SEMS and diverting stoma in relation to an emergency admission 72 hours before the procedures.
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2007-12-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute colorectal cancer surgery (study 1) | At the time of surgery
  Acute surgery as the first surgical intervention for colorectal cancer. This is registered by the surgeon in the DCCG.dk database prior to surgery. A surgical procedure is registered as acute by the surgeon based on clinical symptoms of an abdominal crises and how fast the surgical procedure is performed after onset of acute symptoms.
  There was no defined time limit from onset of symptoms to onset of procedure in order to classify the procedure as acute. This was up to the surgeon who registered the patient.
Postoperative 1-year mortality rate (study 2) | Within 365 days of surgery
  1-year mortality after acute colorectal cancer surgery

SECONDARY OUTCOMES:
Postoperative 90-day mortality (study 2) | Within 90-days of surgery
  90-day mortality after acute colorectal cancer surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thea H. Degett, MD, Principal Investigator — Zealand University Hospital

IPD SHARING:
Plan to Share IPD: No
Since the data belongs to the DCCG.dk database, it is not possible to share them.